CLINICAL TRIAL: NCT05979532
Title: A Longitudinal Prospective, Observational, Cohort Study in Lactating Mothers and Their Newborns to Further Unravel the Complexity of Human Milk
Brief Title: A Study in Lactating Mothers and Their Newborns to Analyse the Composition of Human Milk
Status: Recruiting | Type: Observational
Sponsor: Nutricia Research (Industry)
Responsible Party: Sponsor
Other Study IDs: SBB21R&35943
Record Dates: First submitted 2023-07-31; First posted 2023-08-07 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Breast Feeding; Milk, Human
Keywords: Breast Feeding; Human milk; Research; Lactation; Human Milk Oligosaccharide; HMO
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The samples may be used in future genetic research. Future genetic research on the samples will only be done when the subject has given a separate consent for this.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The current longitudinal (max. 2-year) observational cohort study in 120 lactating mothers and their newborns will make it possible to explore human milk composition across different lactation stages, between different human milk groups, and in relation to maternal, perinatal, infant, and sample characteristics as well as to the microbiota of the infant.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women in the third trimester of pregnancy (≥28 weeks) who have the intention to provide breastfeeding for at least 6 months post-partum.
* Age ≥ 18 years.
* Willingness to provide residual human milk.
* Living in proximity of NCRU (clinical site in NL).
* Dutch speaking and reading.
* Freezer -18°C available.
* Having mobile phone, tablet, or computer available.
* Signed informed consent from the subject (pregnant woman).
* Signed informed consent from the other parent and/or legally acceptable representative, of the unborn baby(s), aged ≥ 18 years.

Exclusion Criteria:

* Pregnant women known positive for human immunodeficiency virus (HIV), hepatitis B (HBV), or hepatitis C (HCV).
* Multiple pregnancy > 2.
* Incapability of subjects to comply with study protocol as per the judgment of the site staff (e.g. fluency in local language, access to laptop/smartphone devices and internet connection required for data collection).
* Women (and their unborn baby(s)) with current or intended participation in any other clinical study involving investigational or marketed products.
* Employees and/or children/family members or relatives of employees of Nutricia Research or the participating site.

Continuation exclusion criteria (after birth)

* Stillbirth
* Newborn having any congenital abnormality, chromosomal disorder or severe disease that would prevent the infant from breastfeeding and/or growing normally based on the opinion of a health care professional and/or study physician.
* No donation of any milk sample within the first 8 weeks postpartum (timepoints week 1, week 1.5, and week 4).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The study population consists of lactating mothers and their newborn.
Study Population: 120 Lactating mothers who have the intention to breastfeed for at least 6 months and their newborns.
Sampling Method: Non-Probability Sample
Enrollment: 172 (Estimated)
Dates: Start 2024-02-13 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Examples of exploratory outcome parameters in this study are the following human milk outcome parameters. | at Day 3 and at Week 1.5, 4, 10, 26, 52, and 104 postpartum.
  Laboratory analyses of Human Milk Oligosaccharides (HMOs), proteins, amino acids, lipids, and fatty acids.
The following exploratory faecal outcome parameter will be analysed if sufficient faecal samples are collected. | at Day 3 and at Week 1.5, 4, 10, 26, 52, and 104 postpartum.
  Laboratory analyses of Infant's faecal microbiome composition.

CONTACTS AND LOCATIONS:
Locations (1):
- Danone Nutricia Research, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No